CLINICAL TRIAL: NCT02150551
Title: Safety and Tolerability Of Allogeneic Mesenchymal Stromal Cells in Pediatric Inflammatory Bowel Disease
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Catherine Bollard (Other)
Responsible Party: Sponsor-Investigator, Catherine Bollard, Director- Center for Emerging Technologies in Immune Cell Therapies (CETI), Children's National Research Institute
Organization: Children's National Research Institute (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: STOMP
Record Dates: First submitted 2014-01-10; First posted 2014-05-30 (Estimated); Results first posted 2023-01-20 (Actual); Last update posted 2024-05-06 (Actual); Status verified 2024-04

CONDITIONS: Inflammatory Bowel Diseases
Keywords: Crohn disease; ulcerative colitis; mesenchymal stromal cells; inflammatory bowel diseases
MeSH Terms: conditions — Inflammatory Bowel Diseases; Crohn Disease; Colitis, Ulcerative

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Mesenchymal Stromal Cells (MSCs) (Experimental): A fixed dose of Mesenchymal Stromal Cells (MSCs) will be studied: 1 x 106 cells/kg administered intravenously (IV) weekly for 4 consecutive weeks, with the option of an additional 4 weeks of treatment, at the discretion of the principal investigator.
  Interventions: Biological: Allogeneic bone marrow-derived mesenchymal stromal cells

INTERVENTIONS:
Biological: Allogeneic bone marrow-derived mesenchymal stromal cells — This study is a pilot phase 1 study of patients with moderately to severely active Crohn Disease (CD) and ulcerative colitis (UC) (≥ 18 years, Mayo score: ≥6 or CDAI: ˃ 220; <18 years, Pediatric Crohn's Disease Activity Index (PCDAI) :> 30) or Pediatric Ulcerative Colitis Activity Index (PUCAI) : >34). A fixed dose will be studied: 1 x 106 cells/kg administered intravenously (IV) weekly for 4 consecutive weeks, with the option of an additional 4 weeks of treatment, at the discretion of the principal investigator.

SUMMARY:
In this trial, investigators will infuse donor bone marrow mesenchymal stromal cells intravenously, as a treatment for pediatric Crohn's disease or ulcerative colitis that has not responded to conventional therapies. The goals of this study are to test the safety and tolerability of donor mesenchymal stromal cells in children with Inflammatory Bowel Disease.

Mesenchymal stromal cells support the development of blood cells within the bone marrow. When isolated from a donor and infused into an animal or human, they have been demonstrated to travel to areas of inflammation, to alter immune responses, to decrease pro-inflammatory cytokines, and to promote tissue repair. Infusion of these cells does not lead to rejection. These properties lead investigators to hypothesize that that these may be they may be beneficial in treating inflammatory bowel disease.

DETAILED DESCRIPTION:
In this trial, investigators will infuse donor bone marrow mesenchymal stromal cells intravenously, as a treatment for pediatric Crohn's disease or ulcerative colitis that has not responded to conventional therapies. Mesenchymal stromal cells support the development of blood cells within the bone marrow. They have also been demonstrated to travel to areas of inflammation, to alter immune responses, to decrease pro-inflammatory cytokines, and to promote tissue repair. Infusion of these cells does not lead to rejection. These properties lead investigators to hypothesize that that these may be they may be beneficial in treating inflammatory bowel disease.

Investigators will culture donated bone marrow mesenchymal stromal cells in a unique automated system, and infuse the cells in a fresh, replicating stage of growth. This study is to test the safety and tolerability of donor mesenchymal stromal cells in children with Inflammatory Bowel Disease.

ELIGIBILITY:
Inclusion Criteria:

* For the young adult cohort, patients must be ages 17 ≤22 years
* For the pediatric cohort, patients must be ages 12 ≤16 years
* Patients must have moderate-severely active CD or UC (defined in section 2.3), and documented active disease on flexible sigmoidoscopy, colonoscopy or MR enterography within the preceding 2 months.
* Patients who have failed or are intolerant of biologic therapy. Specifically, the patient will have recurrence or persistence of active disease despite current or past treatment with a biologic. At the time of enrollment, study subjects may be currently receiving 5-aminosalicylates, corticosteroids (≤ 20 mg daily or up to 0.5 mg/kg/day if weight <40 kg), methotrexate, 6MP/azathioprine, or a biologic (either as monotherapy or in combination). During the treatment phase, if the treating physician thinks that a medication dose should be lowered to avoid side effects, this should be recorded.
* Patient or parent/guardian capable of providing informed consent.

Exclusion Criteria:

* • Patients < 12 years of age or >22 years of age
* Pregnant or breastfeeding. Serum pregnancy test must be negative at screening for female subjects of childbearing potential. Urine pregnancy test must remain negative at each of 4 infusion visits.
* Patients with toxic mega-colon or intestinal perforation
* Evidence of autoimmune chronic active hepatitis or sclerosing cholangitis.
* Patients with fever > 39° C or clinically significant active infection within 1 week (i.e. chronic infections including Hepatitis B/C or HIV or acute infections, including urinary tract infection and respiratory tract infection)
* Received an agent not approved by the FDA for marketed use in any indication or any small molecule inhibitors (i.e. naltrexone) within 60 days of enrollment.
* Subjects who are taking greater than 20 mg (or if body weight <40 kg, 0.5 mg/kg) of prednisone daily.
* Clinically significant abnormal biochemical and hematological parameters, including:

  * Neutrophil count < 1000 cells/mm3
  * Hemoglobin < 8 g/dl
  * Platelet count ≤ 130 cells/mm3
  * Creatinine ≥ 1.2 x the upper limit of normal
  * Alanine aminotransferase (ALT) and/or aspartate aminotransferase (AST) ≥ 2x the upper limit of normal
  * Conjugated bilirubin greater than 1.2. mg/dL
* Has active infection with enteric pathogens as evidenced by positive microbiological culture of stool or C.difficile toxin PCR.
* Had bowel surgery other than perianal procedures (fistulotomy, seton placement, abscess drainage) within 3 months of enrollment.
* Has uveitis
* Has known pulmonary disease, excluding mild intermittent asthma

Ages: 12 Years to 22 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 1 (Actual)
Dates: Start 2018-06-07 (Actual); Primary Completion 2018-09-05 (Actual); Study Completion 2018-09-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Laurie S. Conklin, M.D., Principal Investigator — Children's National Research Institute
Locations (1):
- Children's National Medical Center, Washington D.C., District of Columbia, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: STOMP001 was enrolled in the study on 6/7/2018 at CNH outpatient clinic. Only one patient was enrolled in this study.
Period: Overall Study
Arm/Group | Mesenchymal Stromal Cells (MSCs)
Started | 1
Completed | 1
Not Completed | 0

BASELINE CHARACTERISTICS:
Population: STOMP001 was enrolled in the study on 6/7/2018 and was withdrawn from the study 09/05/2018 due to refusal to continue the follow-up visits for the study.
Arm/Group | Mesenchymal Stromal Cells (MSCs)
Number analyzed (Participants) | 1
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 1
  >=65 years | 0
Age, Customized [Number; unit: years]
  1 | 1
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1
  Male | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 1
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 1

OUTCOME MEASURES:

1. Primary Outcome: Number of Subjects Who Experience Serious Adverse Events, Adverse Events, and/or Early Treatment Discontinuations.
Description: Safety and tolerability of the administration of human allogeneic bone marrow-derived stromal cells to children and young adults with IBD, measured by the frequency of any SAEs, AEs and/or early treatment discontinuations. Weekly infusions for 8 weeks, post-treatment assessment 45 days after last infusion, three additional follow-up visits over 2 years.
Time Frame: 45 days after the last infusion
Population: STOMP001 was enrolled in the study on 6/7/2018 and was withdrawn from the study 09/05/2018 due to refusal to continue the follow-up visits for the study. Due to patient's refusal to continue the study, there were no relative data to be analyzed.
Measure: Count of Participants; unit: Participants
Arm/Group | Mesenchymal Stromal Cells (MSCs)
Number analyzed (Participants) | 1
Participants | 1

2. Secondary Outcome: Proportion of Patients With Clinical Response
Description: Proportion of subjects that achieve a clinical response by 45 days after last infusion, as defined by a decrease in PCDAI from baseline by greater than or equal to 12.5 points (for CD) or a decrease in PUCAI of greater than or equal to 20 points (for UC).
Time Frame: 45 days after last infusion
Population: as for outcome 1
Arm/Group | Mesenchymal Stromal Cells (MSCs)
Number analyzed (Participants) | 0

3. Secondary Outcome: Number of Subjects Demonstrating an Improvement of Laboratory Tests Reflecting Systemic Inflammation.
Description: Improvement in laboratory parameters (i.e. C-reactive protein, fecal calprotectin, anti-HLA antibodies, and viral specific T-cell activity)
Time Frame: 45 days after last infusion
Population: as for outcome 1
Arm/Group | Mesenchymal Stromal Cells (MSCs)
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Time Frame: 3 months
Description: Participant was withdrawn from the study after 3 months due to refusal to continue all study related follow-up visits.
Arm/Group | Mesenchymal Stromal Cells (MSCs)
All-Cause Mortality (participants affected / at risk) | 0/1
Serious Adverse Events (participants affected / at risk) | 1/1
Other Adverse Events (participants affected / at risk) | 1/1
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Mesenchymal Stromal Cells (MSCs) (N=1)
Worsening Crohn's disease (Gastrointestinal disorders) | 1 (1) — On 6/26/2018, patient went to the ER for vomiting and dehydration. Patient was then hospitalized at CNMC on 6/29/18 for conditions consistent with worsening Crohn's disease.
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Mesenchymal Stromal Cells (MSCs) (N=1)
Fainting (Cardiac disorders) | 1 (1) — On 6/11/2018, patient fainted at work and per PI's recommendation, patient went to the ER for labs, EKG and IV fluids
Superior mesenteric artery syndrome (Partial Obstruction of Duodenum) (Gastrointestinal disorders) | 1 (1) — On 6/30/2018, patient developed Superior mesenteric artery syndrome (Partial Obstruction of Duodenum). The event ended on 9/5/2018

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol (2018-01-22): https://cdn.clinicaltrials.gov/large-docs/51/NCT02150551/Prot_000.pdf